CLINICAL TRIAL: NCT03679676
Title: Phase 2 Randomized Controlled Trial Using Biologics to Improve Multi OIT Outcomes
Brief Title: Clinical Study Using Biologics to Improve Multi OIT Outcomes (COMBINE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Food Allergy Research & Education (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Medical Director, Clinical Research Unit, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-47935; 5U19AI104209-07 (NIH)
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Hypersensitivity; Food Allergy; Hypersensitivity, Food; Peanut Hypersensitivity; Peanut Allergy
Keywords: Food Allergy; Hypersensitivity, Peanut; Food Hypersensitivity; Allergy, Food
MeSH Terms: conditions — Hypersensitivity; Food Hypersensitivity; Peanut Hypersensitivity | interventions — Omalizumab; dupilumab

STUDY DESIGN:
Intervention Model Description: This is a prospective Phase 2, single-center, multi-allergen OIT in participants with proven allergies to 2 or 3 different foods in which one must be peanut. Our intent to treat population will be 110 participants, ages 4 to 55 years with a history of multiple food allergies of 2 or 3 different foods including peanut. Allergy will be confirmed by FA-specific IgE levels and positive skin prick test (SPT). Enrolled participants must be positive during the DBPCFCs at or before the 300 mg (444 mg cumulative) dosing level of FA proteins.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Omalizumab (Other): Participants will be treated with omalizumab for 8 weeks, followed by 24 weeks of treatment with placebo
  Interventions: Drug: Omalizumab; Other: Placebo
- Cohort B: Omalizumab/Dupilumab (Other): Participants will be treated with omalizumab for 8 weeks, followed by 24 weeks of treatment with dupilumab.
  Interventions: Drug: Omalizumab; Drug: Dupilumab
- Cohort C: Dupilumab (Other): Participants will be treated with placebo for 8 weeks, followed by 24 weeks of treatment with dupilumab.
  Interventions: Drug: Dupilumab; Other: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab is injected every 2 to 4 weeks
  Other Names: Xolair
  Arms: Cohort A: Omalizumab; Cohort B: Omalizumab/Dupilumab
Drug: Dupilumab — Dupilumab is injected every 2 weeks
  combination, or placebo.
  Other Names: Dupixent
  Arms: Cohort B: Omalizumab/Dupilumab; Cohort C: Dupilumab
Other: Placebo — Placebo is injected every 2 to 4 weeks
  Arms: Cohort A: Omalizumab; Cohort C: Dupilumab

SUMMARY:
Food allergy (FA) is a serious public health concern that causes potentially-life threatening reactions in affected patients. The prevalence of food allergy in the United States (U.S.) has increased substantially and now affects 15 million patients:4-8% of children (6 million children, 30% with multiple food allergies) and about 9% of adults. This is a prospective Phase 2, single-center, multi-allergen OIT study in participants with proven allergies to 2 or 3 different foods in which one must be a peanut. The total of participants in the clinical study will be 110, ages 4 to 55 years with a history of multiple food allergies of 2 to 3 different foods including peanut. Allergy will be confirmed by FA-specific IgE levels and positive skin prick test (SPT). Enrolled participants must be positive during the Double-blind Placebo-controlled Food challenge (DBPCFC) at or before the 300 mg (444 mg cumulative) dosing level of FA proteins.

DETAILED DESCRIPTION:
This is a prospective Phase 2, single-center, multi-allergen OIT study in participants with proven allergies to 2 or 3 different foods in which one must be peanut. The total population will be 110 participants, ages 4 to 55 years that present with a history of multiple food allergies of 2 or 3 different foods including peanut, food-allergen (FA)-specific IgE levels, and positive skin prick test (SPT).

Enrolled participants must react positively during DBPCFCs at or before the 300 mg (444 mg cumulative) dosing level of FA proteins of 2 or 3 allergens in which one must be a peanut.

There will be three study cohorts, all will be double blinded:

Cohort A (50 participants) will be treated with omalizumab for 8 weeks followed by 24 weeks of treatment with placebo. Cohort B (50 participants) will be treated with omalizumab for 8 weeks, followed by 24 weeks of treatment with dupilumab. Cohort C (10 participants) will be treated with placebo for 8 weeks followed by 24 weeks treatment with dupilumab. All cohorts will receive multifood allergen oral immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 through 55 years (inclusive).
* Clinical history of peanut allergy and 1 or 2 additional foods from the following foods: milk, almond, shellfish, fish, cashew, hazelnut, egg, walnut, sesame seeds, soy, and wheat. Allergy to milk and egg is defined as unable to tolerate both cooked and uncooked forms.
* Positive allergy test determined by:
* ImmunoCAP serum IgE level >4 kUA/L for each allergen within the past 12 months OR
* Skin prick test (SPT) ≥6 mm wheal diameter to each allergen.
* A clinical reaction during a DBPCFC to small doses of food defined as a cumulative dose of =/<444 mg food protein.
* No clinical reaction observed during the placebo (oat) challenge.
* Subject and/or parent guardian must be able to understand and provide informed consent.
* Written informed consent from adult participants.
* Written informed consent from parent/guardian for minor participants.
* Written assent from minor participants as appropriate (e.g., at and above the age of 7 years).
* Use of effective birth control by female participants of childbearing potential.

Exclusion Criteria:

* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension.
* Individuals less than 15 kg in weight at start of the study
* History of severe anaphylaxis to participant-specific foods that will be used in this study, defined as neurological compromise or requiring intubation.
* History of chronic disease (other than asthma, atopic dermatitis or allergic rhinitis) that is, or is at significant risk of becoming, unstable or requiring a change in chronic therapeutic regimen.
* History of eosinophilic esophagitis (EoE), another eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia (e.g., difficulty swallowing, food "getting stuck"), or recurrent gastrointestinal symptoms of undiagnosed etiology.
* Severe asthma (NAEPP EPR-3 Medication Criteria Steps 5 or 6)
* Mild or moderate asthma (NAEPP EPR-3 Medication Criteria Steps 1-4), if uncontrolled or difficult to control.
* Uncontrolled asthma as evidenced by:

  * FEV1 < 80% of predicted, or ratio of FEV1 to forced vital capacity (FEV1/FVC) < 75% of predicted, with or without controller medications (only for age 6 or greater and able to do spirometry reliably. If unable to do spirometry, PEF of >80% is acceptable) or;
  * One overnight admission to a hospital in the past year for asthma or;
  * Emergency room (ER) visit for asthma within six months prior to screening.
* Inability to tolerate biological (antibody) therapies.
* Use of immunomodulator therapy (not including corticosteroids).
* Use of beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers.
* Current participation or within the last 4 months in any other interventional study.
* Pregnancy or lactation.
* Allergy to oat (placebo in DBPCFC).
* Use of investigational drugs within 16 weeks of participation.
* In build up phase of immunotherapy for aeroallergens or venom.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
The success rates of passing a peanut Double-Blind Placebo Controlled Food Challenge (DBPCFC) | 44 weeks
  Success is defined as passing a cumulative dose of >=1,043 mg at the Week 44 DBPCFC if the subject has no or mild objective reactions. The primary endpoints would be compared between cohort A and cohort B.
The success rates of passing a DBPCFC to peanut and at least one other FA | 44 weeks
  Success is defined as passing a cumulative dose of >=1,043 mg at the Week 44 DBPCFC if the subject has no or mild objective reactions. The primary endpoints would be compared between cohort A and cohort B.
The success rates of passing a DBPCFC to peanut and two other FAs | 44 weeks
  Success is defined as passing a cumulative dose of >=1,043 mg at the Week 44 DBPCFC if the subject has no or mild objective reactions. The primary endpoints would be compared between cohort A and cohort B.

SECONDARY OUTCOMES:
Proportion of participants who successfully pass DBPCFCs to a cumulative dose of >=1,043 mg protein to 1, 2, or 3 FAs when applicable at week 44 | 44 weeks
Proportion of participants who successfully pass DBPCFCs to a cumulative dose of ≥2,043 mg to 1, 2, or 3 FAs when applicable at week 32 | 32 weeks
Proportion of participants who pass DBPCFCs for each FA at a cumulative dose of ≥1,043 mg, ≥2,043 mg, or ≥4,043 mg at week 32 and/or week 44. | week 32 and/or 44
Proportion of participants who have a 10-fold change in the cumulative tolerance dose for each FA at weeks 32 and/or week 44, compared to baseline | Baseline and week 32 and/or 44

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca S Chinthrajah, M.D., Study Director — Sean N Parker Center for Allergy and Asthma Center at Stanford
Locations (3):
- United States (3):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Sean N. Parker Center for Allergy & Asthma Research at Stanford University, Palo Alto, California
  - University of California San Diego (UCSD), San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736
- See also: Related Info — http://med.stanford.edu/allergyandasthma/clinical-trials.html

DOCUMENTS (1):
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03679676/ICF_000.pdf